CLINICAL TRIAL: NCT03071354
Title: Phase II, Multi-center, Randomized Control Trial of Beta- Hydroxy-Methyl-Butyrate (HMB) in Improving Physical Muscle Function, in Nutritionally at Risk, Elderly Patients
Brief Title: Improving Muscle Function in Nutritionally at Risk, Elderly Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is Moving Institutions
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00035962
Record Dates: First submitted 2017-02-28; First posted 2017-03-06 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-08

CONDITIONS: Muscle Weakness; ICU-acquired Weakness
Keywords: ICU-acquired weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMB Protein Supplementation Group (Experimental): Intervention patients will receive 2 x 237mL bottles of the commercially available liquid HMB protein supplement (3g) (Ensure Active™ Muscle Health) throughout the study.
  In addition, all patients will be fed according to the Canadian Critical Nutrition Practice Guidelines, and protein/energy requirements will be determined by the local dietitians according to their local practice standards.
  Interventions: Dietary Supplement: HMB protein supplement (3g)
- Control Group (Active Comparator): Control patients will receive 2 x 237mL bottles of the commercially available nutritional supplement (Ensure® Original) throughout the study.
  In addition, all patients will be fed according to the Canadian Critical Nutrition Practice Guidelines, and protein/energy requirements will be determined by the local dietitians according to their local practice standards.
  Interventions: Dietary Supplement: Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: HMB protein supplement (3g) — HMB 3g/day or iso-nitrogenous control (discussed below) in addition to standard enteral, and parenteral nutritional supplementation and standard nutrition when transferred to the ward. The dose of HMB was chosen based on multiple studies revealing efficacy of 3g/day improving muscle mass and demonstrating an excellent safety profile. Feeding will be initiated as per local practice. Enrolled patients will be randomized to supplementation with HMB (3g) or control will begin within 72 hours of admission to ICU.
  Other Names: Ensure Active™ Muscle Health
  Arms: HMB Protein Supplementation Group
Dietary Supplement: Nutritional Supplement — Control patients will receive 2 x 237mL bottles of the commercially available nutritional supplement (Ensure® Original) in addition to standard enteral, and parenteral nutritional supplementation and standard nutrition when transferred to the ward throughout the study. While the patient is intubated, the control nutritional supplement will be delivered via the enteral feeding tube. The participant will switch to oral administration once extubated
  Other Names: Ensure® Original
  Arms: Control Group

SUMMARY:
The investigators propose to conduct a randomized, control trial of β-hydroxy-β-methylbutyrate (HMB) supplementation in elderly patients (≥65 years of age) with acute respiratory failure, who are identified at high risk for malnutrition by ICU-specific nutritional risk scores. Patients will receive either 3g of HMB daily, or control, daily until day 28 following randomization (even if discharged).The investigators will measure functional outcomes using standard, validated measures prior and after discharge.

DETAILED DESCRIPTION:
The investigators propose to conduct a randomized, control trial of HMB supplementation in elderly patients (≥65 years of age) with acute respiratory failure, who are identified at high risk for malnutrition by ICU-specific nutritional risk scores. Patients will receive either 3g of HMB daily, or control, daily until day 28 following randomization (even if discharged).the investigators will measure functional outcomes using standard, validated measures prior and after discharge.

The investigators hypothesize that this inexpensive nutrient, HMB, along with our supportive measures, reduces muscle loss, improves physical muscle function, and improves quality of life in the longer term following critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age ≥65 years.
2. Acute respiratory failure (ARF, defined by expected mechanical ventilation for > 72 hours from the point of screening)
3. Elevated nutritional risk (NUTRIC score>5 - see below).

Exclusion Criteria:

1. Over 72 hours from ICU admission.
2. Not expected to survive another 48 hours
3. Lack of commitment to full, aggressive care
4. Patients who have an absolute contraindication to EN (obstruction, perforation, high output fistula),
5. Pregnant women
6. Prisoners
7. Known allergy to study nutrients
8. Unable to walk prior to current illness.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance | At 42 days follow up
  Maximum distance walked by subject in 6 minutes on level ground

SECONDARY OUTCOMES:
Body Composition-Calf circumference | At 42 days follow up
  Measurement of the calf circumference
Body Composition-Quadriceps layer muscle thickness (QLMT) | At 42 days follow up
  Thigh ultrasound for quadriceps muscle thickness
Hand-grip strength (HGS) | At 42 days follow up
  Measurement of force of isometric grip strength using hand-held dynamometer
Timed Get Up and Go test | At 42 days follow up
  Time for subject to go from sitting to standing unaided

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Agarwala, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided